CLINICAL TRIAL: NCT01437995
Title: Long-acting Beta Agonist Step Down Study
Acronym: LASST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: American Lung Association (Other); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Robert A. Wise, Professor of Medicine, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ADV115922
Record Dates: First submitted 2011-09-05; First posted 2011-09-21 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-03

CONDITIONS: Asthma
Keywords: Asthma; Step down therapy; Inhaled corticosteroids; Long-acting beta agonists; Fluticasone Salmeterol
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Salmeterol Xinafoate; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fluticasone/Salmeterol Diskus 250/50 ug (Active Comparator): Continuation of Fluticasone/Salmeterol Diskus 250/50 ug twice daily
  Interventions: Drug: Fluticasone/Salmeterol Diskus
- Fluticasone/Salmeterol Diskus 100/50 ug (Active Comparator): Reduced dose Fluticasone/Salmeterol Diskus 100/50 ug twice daily
  Interventions: Drug: Fluticasone/Salmeterol Diskus
- Fluticasone Diskus alone 250 ug (Active Comparator): Fluticasone Diskus alone 250 ug twice daily without Salmeterol
  Interventions: Drug: Fluticasone Diskus

INTERVENTIONS:
Drug: Fluticasone/Salmeterol Diskus — Continuation of Fluticasone/Salmeterol Diskus 250/50 ug twice daily
  Other Names: Fluticasone; Salmeterol
  Arms: Fluticasone/Salmeterol Diskus 250/50 ug
Drug: Fluticasone/Salmeterol Diskus — Reduced dose Fluticasone/Salmeterol Diskus 100/50 ug twice daily
  Other Names: Fluticasone; Salmeterol
  Arms: Fluticasone/Salmeterol Diskus 100/50 ug
Drug: Fluticasone Diskus — Fluticasone Diskus alone 250 ug twice daily without Salmeterol
  Other Names: Fluticasone
  Arms: Fluticasone Diskus alone 250 ug

SUMMARY:
This study is a 56-week, multi-center, blinded, randomized, double-masked parallel group comparative effectiveness study of approaches to stepping down therapy for patients with well-controlled asthma treated with combination ICS and LABA.

DETAILED DESCRIPTION:
Current asthma guidelines recommend stepping down therapy once asthma is controlled for at least 3 months. For patients treated with inhaled corticosteroids (ICS) alone, a dose reduction of 25-50% to a minimal dose that controls disease is recommended. The optimal approach to reducing treatment in patients with asthma treated with combination inhaled corticosteroids and long-acting beta agonists (ICS/LABA) is not clear. The American Lung Association Asthma Clinical Research Center (ALAACRC) is a network of 18 asthma research centers with the goal of performing clinical trials directly relevant to clinical practice. The question of the optimal way to de-escalate therapy in patients with asthma that is well controlled on fixed dose combination ICS/LABA is a key question for practitioners caring for patients with moderate to severe persistent asthma. We propose a 56 week multi-center, prospective, randomized, three-arm parallel group comparative effectiveness study comparing three approaches to care of patients with asthma well-controlled for three months on combination ICS/LABA: reduction of ICS dose and maintenance of LABA, initial discontinuation of LABA with continuation of ICS, and continuation of stable dose ICS/LABA. Our primary goal is to perform a pragmatic study that resembles clinical practice and determine the optimal treatment strategy that results in the lowest rate of treatment failure over 48 weeks of follow-up. Additional exploratory analyses include assessing risk factors for step-down failure, and to assess the duration of time that asthma control is maintained when therapy is de-escalated.

ELIGIBILITY:
Inclusion Criteria:

* age 12-80 years
* physician diagnosed asthma that is well-controlled on moderate dose ICS/LABA based on an Asthma Control Test (ACT) score more than or equal to 20, and the absence of unscheduled visits or use of rescue prednisone for 4 weeks prior to enrollment
* pre-bronchodilator FEV1 (forced expiratory volume in 1 second) more than or equal to 70% predicted

Exclusion Criteria:

* chronic oral steroid therapy
* hospitalization or urgent care visit within 4 weeks of the screening visit
* lung disease other than asthma including COPD, bronchiectasis, sarcoidosis or other lung disease
* less than 10 pack/yr of tobacco use and abstinence for at least 1 yr
* history of extensive environmental tobacco exposure or occupational exposure suggestive of possible COPD (chronic obstructive pulmonary disease) per judgment of investigator
* post bronchodilator FEV1 less than 70% predicted
* near fatal asthma (intubation or ICU admission for asthma) within 2 yrs of enrollment
* high risk of near fatal or fatal asthma
* history of known premature birth less than 33 weeks or any significant level of respiratory care including prolonged oxygen administration or mechanical ventilation during the neonatal period
* unstable cardiac disease (decompensated congestive heart failure, unstable angina, recent myocardial infarction, atrial fibrillation, supraventricular or ventricular tachycardia, congenital heart disease, or severe uncontrolled hypertension)
* other major chronic illnesses which in the judgment of the study physician would interfere with participation in the study e.g. including but not limited to uncontrolled diabetes, uncontrolled HIV infection or other immune system disorder
* drug allergies to any component of study drug or history of adverse reaction to short or long acting beta agonists
* for women of child bearing potential; not pregnant, not lactating and agree to practice an adequate birth control method (abstinence, combination barrier and spermicide, or hormonal) for the duration of the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2012-03; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Wise, MD, Study Director — Johns Hopkins University; Linda Rogers, MD, Principal Investigator — NYU Langone Health
Locations (19):
- United States (19):
  - University of Arizona, Arizona Respiratory Center, Tucson, Arizona
  - University of California, San Diego, San Diego, California
  - National Jewish Health, Denver, Colorado
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami/University of South Florida, Tampa, Florida
  - The Illinois Consortium, Chicago, Illinois
  - St. Vincent Healthcare, Indianapolis, Indiana
  - St. Vincent Hospital and Health Care Center, Inc, Indianapolis, Indiana
  - Louisiana State University Health Sciences Center, The Ernest N. Morial Asthma, Allergy and Respiratory Disease Center, New Orleans, Louisiana
  - University of Missouri, Kansas City School of Medicine, Kansas City, Missouri
  - Washington University/St. Louis University, St Louis, Missouri
  - Hofstra North Shore-LIJ School of Medicine, New Hyde Park, New York
  - New York University School of Medicine, New York, New York
  - Maria Fareri Children's Hospital at Westchester Medical Center and New York Medical College, Valhalla, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Ohio State University Medical Center, Columbus, Ohio
  - Baylor College of Medicine, Houston, Texas
  - Northern New England Consortium, Colchester, Vermont
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Derived] Blake KV, Antal H, Bunnell HT, He J, Henderson R, Holbrook JT, McCahan SM, Pennington C, Rogers L, Shade D, Sugar EA, Taylor A, Wise RA, Wysocki T. Comprehension by Caregivers and Adolescents of Clinical Trial Information Delivered via Multimedia Video Versus Conventional Practice: Nonrandomized Controlled Trial. JMIR Pediatr Parent. 2023 Jun 22;6:e44252. doi: 10.2196/44252. PMID 37347518
- [Derived] DiMango E, Rogers L, Reibman J, Gerald LB, Brown M, Sugar EA, Henderson R, Holbrook JT. Risk Factors for Asthma Exacerbation and Treatment Failure in Adults and Adolescents with Well-controlled Asthma during Continuation and Step-Down Therapy. Ann Am Thorac Soc. 2018 Aug;15(8):955-961. doi: 10.1513/AnnalsATS.201711-886OC. PMID 29863899
- See also: American Lung Association — http://www.lungusa.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled participants were enrolled in an 8-week open label treatment run-in and were subsequently randomized only if their asthma remained stable (i.e. an ACT score ≥ 20 at weeks 4 & 8, no unscheduled healthcare encounters, no change in asthma medication, pre-bronchodilator FEV1 ≥ 70% predicted, and limited use of rescue beta-agonist).
Groups:
- Stable ICS-LABA: Continuation of Fluticasone/Salmeterol Diskus 250/50 ug twice daily
  Fluticasone/Salmeterol Diskus: Continuation of Fluticasone/Salmeterol Diskus 250/50 ug twice daily
- Reduced ICS/LABA: Reduced dose Fluticasone/Salmeterol Diskus 100/50 ug twice daily
  Fluticasone/Salmeterol Diskus: Reduced dose Fluticasone/Salmeterol Diskus 100/50 ug twice daily
- LABA Step Off: Fluticasone Diskus alone 250 ug twice daily without Salmeterol
  Fluticasone Diskus: Fluticasone Diskus alone 250 ug twice daily without Salmeterol
Period: Overall Study
Arm/Group | Stable ICS-LABA | Reduced ICS/LABA | LABA Step Off
Started | 151 | 149 | 155
Included in Treatment Failure Analysis | 150 | 146 | 151
Completed | 140 | 131 | 135
Not Completed | 11 | 18 | 20
Not completed — Lost to Follow-up | 11 | 18 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stable ICS-LABA | Reduced ICS/LABA | LABA Step Off | Total
Number analyzed (Participants) | 151 | 149 | 155 | 455
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [22 to 51] | 33 [17 to 49] | 35 [23 to 50] | 35 [20 to 50]
Age, Customized [Number; unit: participants]
  <18 | 31 | 39 | 30 | 100
  >=18 | 120 | 110 | 125 | 355
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 88 | 103 | 287
  Male | 55 | 61 | 52 | 168
Race/Ethnicity, Customized [Number; unit: participants]
  White | 72 | 74 | 75 | 221
  Black | 52 | 48 | 51 | 151
  Hispanic | 19 | 23 | 24 | 66
  Other | 8 | 4 | 5 | 17
Region of Enrollment [Number; unit: participants]
  United States | 151 | 149 | 155 | 455
Smoke exposure [Number; unit: participants] — History of cigarette smoking and current exposure to secondhand smoke. Individuals with no history of cigarette smoking and no current exposure to second hand smoke are not counted.
  participants
    Former smoker | 23 | 25 | 14 | 62
    Secondhand smoke home/work | 18 | 21 | 17 | 56
Asthma characteristics [Number; unit: participants] — Description of characteristics of recent asthma treatment. Individuals who did not have a history of the treatment were not counted.
  participants
    Hospitalized for asthma in past year | 5 | 3 | 6 | 14
    Oral steroids in past year | 44 | 36 | 42 | 122
    Daily short-acting beta agonist use | 7 | 12 | 10 | 29
    Daily anti-leukotriene use | 32 | 30 | 30 | 92
Age of Asthma Onset [Median (Inter-Quartile Range); unit: years] | 7 [3 to 21] | 7 [2 to 18] | 7 [2 to 20] | 7 [2 to 20]
eNO (exhaled nitric oxide) [Median (Inter-Quartile Range); unit: parts per billion] | 18.5 [12.5 to 26.5] | 17.5 [13.8 to 25.3] | 16.5 [11.5 to 26.5] | 17.5 [12.5 to 26]
Atopy (phadiatop ≥ 0.35 kUA/l) [Number; unit: participants] | 115 | 123 | 114 | 352
Asthma Symptom Utility Index [Median (Inter-Quartile Range); unit: units on a scale] — The Asthma Symptom Utility Index asks about asthma symptoms within the past 2 weeks. The scale ranges from 0 to 1 with higher scores indicating better health.
  units on a scale | 0.95 [0.90 to 1.00] | 0.94 [0.89 to 1.00] | 0.98 [0.92 to 1.00] | 0.95 [0.89 to 1.00]
Pulmonary function measures [Median (Inter-Quartile Range); unit: Liters]
  Pre-bronchodilator FEV1 | 2.82 [2.24 to 3.31] | 2.86 [2.35 to 3.44] | 2.82 [2.38 to 3.49] | 2.83 [2.30 to 3.43]
  Pre-bronchodilator FVC | 3.54 [2.99 to 4.30] | 3.62 [2.97 to 4.54] | 3.65 [3.03 to 4.56] | 3.62 [3.00 to 4.44]
  Post-bronchodilator FEV1 | 2.88 [2.34 to 3.36] | 2.96 [2.39 to 3.50] | 2.93 [2.44 to 3.60] | 2.92 [2.39 to 3.49]
  Post-bronchodilator FVC | 3.59 [3.09 to 4.28] | 3.72 [3.11 to 4.63] | 3.65 [3.06 to 4.52] | 3.62 [3.09 to 4.50]
Pulmonary function measures, percent predicted [Median (Inter-Quartile Range); unit: percent predicted]
  Pre-bronchodilator FEV1 | 91 [82 to 99] | 91 [83 to 101] | 92 [83 to 101] | 91 [83 to 101]
  Pre-bronchodilator FVC | 98 [89 to 107] | 100 [91 to 107] | 98 [90 to 108] | 99 [90 to 107]
  Pre-bronchodilator peak flow | 96 [84 to 110] | 100 [90 to 110] | 98 [89 to 113] | 98 [88 to 110]
Other conditions, based upon self-report [Number; unit: participants]
  Eczema | 35 | 28 | 26 | 89
  Sinusitis | 50 | 41 | 34 | 125
  Allergic rhinitis | 85 | 73 | 88 | 246
  Food allergies | 33 | 40 | 34 | 107
  Allergies worsen asthma | 123 | 113 | 122 | 358
Pre-bronchodilator peak flow [Median (Inter-Quartile Range); unit: Liters per minute] | 420 [350 to 500] | 430 [350 to 500] | 430 [360 to 500] | 430 [350 to 500]
Asthma Control Test Score [Median (Inter-Quartile Range); unit: units on a scale] — The Asthma Control Test is a validated self-administered survey utilizing 5 questions to assess asthma control on a scale from 1 (poor control) to 5 (total control) in individuals 12 years and older. By answering all 5 questions a patient with asthma can obtain a score that may range between 5 and 25. Asthma control is considered a good characteristic for a person with asthma and therefore a higher score is considered a better outcome.
  units on a scale | 23 [22 to 25] | 23 [21 to 24] | 23 [22 to 24] | 23 [22 to 25]
Marks AQLQ [Median (Inter-Quartile Range); unit: units on a scale] — Marks Asthma Quality of Life Questionnaire (AQLQ) measures physical and emotional asthma specific quality of life during the past four weeks. The minimum score is 0 and the maximum score is 80, with lower scores indicating better quality of life. The scale is for use in adults only (individuals aged 18 or older). Population: The Marks AQLQ is for adults only and was only administered to adult participants (individuals age 18 or older).
  units on a scale
    number analyzed (Participants) | 120 | 110 | 125 | 355
    (all) | 4.0 [1.5 to 8.0] | 5.0 [2.0 to 9.0] | 4.0 [2.0 to 7.0] | 4.0 [2.0 to 8.0]
Children's Health Survey for Asthma - Child Version [Median (Inter-Quartile Range); unit: units on a scale] — The Children's Health Survey for Asthma - Child Version (CHSA-C) is a self-reported measure of functional impairments that are most troublesome to children 12 to 17 years of age as a results of their asthma over the past three weeks. Results are reported in Physical, Activity, and Emotion domains. For all domains, the minimum value is 0 and the maximum value is 100, with higher values indicating better health or more positive outcomes. Population: The Children's Health Survey for Asthma - Child Version (CHSA-C) is for use in individuals under the age of 18 only. The CHSA-C was administered only to those participants under the age of 18 in our study.
  units on a scale
    Physical: number analyzed (Participants) | 31 | 39 | 30 | 100
    Physical | 93 [93 to 100] | 93 [89 to 100] | 96 [93 to 100] | 93 [91 to 100]
    Activity: number analyzed (Participants) | 31 | 39 | 30 | 100
    Activity | 100 [92 to 100] | 100 [92 to 100] | 100 [96 to 100] | 100 [92 to 100]
    Emotional: number analyzed (Participants) | 31 | 39 | 30 | 100
    Emotional | 93 [86 to 98] | 95 [91 to 100] | 93 [88 to 100] | 93 [89 to 100]
Euroqual EQ-5D-5L [Median (Inter-Quartile Range); unit: units on a scale] — The Euroqual EQ-5D-5L is a self-completed generic instrument for measuring quality of life over five dimensions - mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The minimum score is 0 and the maximum score is 1, with higher scores indicating better quality of life or better health state.
  units on a scale | 1.00 [0.86 to 1.00] | 1.00 [0.86 to 1.00] | 1.00 [0.86 to 1.00] | 1.00 [0.86 to 1.00]

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failure
Description: Rate of treatment failures assessed by decline in peak flow or FEV1, increased need for beta agonists, requirement for non-scheduled medical care for asthma symptoms, or prednisone taper.
Time Frame: 48 weeks
Measure: Number; unit: participants
Arm/Group | Stable ICS-LABA | Reduced ICS/LABA | LABA Step Off
Number analyzed (Participants) | 150 | 146 | 151
participants | 38 | 39 | 45
Statistical Analysis 1: Comparison: Stable ICS-LABA vs Reduced ICS/LABA vs LABA Step Off; Test type: Superiority or Other; Hazard Ratio (HR) = 1.07, 95.3% CI 2-sided [0.69 to 1.65]

2. Secondary Outcome: Pulmonary Function- Change in Peak Expiratory Flow
Description: Change in morning peak expiratory flow rate from the patients' daily diary cards, calculated at 48 weeks minus baseline (randomization)
Time Frame: Baseline and 48 weeks
Measure: Median (95% Confidence Interval); unit: Liters per minute
Arm/Group | Stable ICS-LABA | Reduced ICS/LABA | LABA Step Off
Number analyzed (Participants) | 150 | 146 | 151
Liters per minute | -0.08 [-8.10 to 7.94] | 4.40 [-3.46 to 12.26] | -14.16 [-23.1 to -5.22]
Statistical Analysis 1: Comparison: Stable ICS-LABA vs Reduced ICS/LABA; Test type: Superiority or Other; p = 0.43, Kruskal-Wallis
Statistical Analysis 2: Comparison: Stable ICS-LABA vs LABA Step Off; Test type: Superiority or Other; p = 0.022, Kruskal-Wallis
Statistical Analysis 3: Comparison: Reduced ICS/LABA vs LABA Step Off; Test type: Superiority or Other; p = 0.002, Kruskal-Wallis

3. Secondary Outcome: Rate of Episodes of Poor Asthma Control
Description: Rate of episodes of poor asthma control (EPAC) defined by unscheduled medical care, hospitalization, use of oral corticosteroids and/or increased use of rescue medications and/or decrease of 30% or more in morning peak expiratory flow rate
Time Frame: 48 weeks
Measure: Number; unit: Episodes of poor asthma control
Arm/Group | Stable ICS-LABA | Reduced ICS/LABA | LABA Step Off
Number analyzed (Participants) | 152 | 147 | 153
Episodes of poor asthma control | 183 | 164 | 219
Statistical Analysis 1: Comparison: Stable ICS-LABA vs Reduced ICS/LABA; Test type: Superiority or Other; Risk Ratio (RR) = 0.93, 95% CI 2-sided [0.63 to 1.41]
Statistical Analysis 2: Comparison: Stable ICS-LABA vs LABA Step Off; Test type: Superiority or Other; Risk Ratio (RR) = 1.18, 95% CI 2-sided [0.80 to 1.73]
Statistical Analysis 3: Comparison: Reduced ICS/LABA vs LABA Step Off; Test type: Superiority or Other; Risk Ratio (RR) = 1.24, 95% CI 2-sided [0.83 to 1.81]

4. Secondary Outcome: Change in Pulmonary Function: FEV1 and FVC
Description: Change in participant's pre-bronchodilator pulmonary function tests (FEV1 and FVC) calculated as 48 weeks minus baseline.
Time Frame: Baseline and 48 weeks
Measure: Median (95% Confidence Interval); unit: Liters
Arm/Group | Stable ICS-LABA | Reduced ICS/LABA | LABA Step Off
Number analyzed (Participants) | 150 | 146 | 151
Liters
  Pre-bronchodilator FEV1 | -0.02 [-0.07 to 0.03] | -0.07 [-0.12 to -0.01] | -0.13 [-0.18 to -0.09]
  Pre-bronchodilator FVC | -0.01 [-0.06 to 0.04] | -0.04 [-0.10 to 0.01] | -0.09 [-0.14 to -0.03]
Statistical Analysis 1: Comparison: Stable ICS-LABA vs Reduced ICS/LABA; Comparing change in pre-bronchodilator FEV1; Test type: Superiority or Other; p = 0.15, Kruskal-Wallis
Statistical Analysis 2: Comparison: Stable ICS-LABA vs LABA Step Off; Comparing change in pre-bronchodilator FEV1; Test type: Superiority or Other; p < 0.001, Kruskal-Wallis
Statistical Analysis 3: Comparison: Reduced ICS/LABA vs LABA Step Off; Comparing change in pre-bronchodilator FEV1; Test type: Superiority or Other; p = 0.027, Kruskal-Wallis
Statistical Analysis 4: Comparison: Stable ICS-LABA vs Reduced ICS/LABA; Comparison of change in pre-bronchodilator FVC; Test type: Superiority or Other; p = 0.40, Kruskal-Wallis
Statistical Analysis 5: Comparison: Stable ICS-LABA vs LABA Step Off; Comparison of change in pre-bronchodilator FVC; Test type: Superiority or Other; p = 0.032, Kruskal-Wallis
Statistical Analysis 6: Comparison: Reduced ICS/LABA vs LABA Step Off; Comparison of change in pre-bronchodilator FVC; Test type: Superiority or Other; p = 0.21, Kruskal-Wallis

5. Secondary Outcome: Pulmonary Function: Change in FEV1/FVC Ratio
Description: Change in participant's FEV1/FVC ratio calculated as 48 weeks minus baseline.
Time Frame: Baseline and 48 weeks
Measure: Median (95% Confidence Interval); unit: ratio
Arm/Group | Stable ICS-LABA | Reduced ICS/LABA | LABA Step Off
Number analyzed (Participants) | 150 | 146 | 151
ratio | -0.002 [-0.009 to 0.005] | -0.009 [-0.016 to -0.002] | -0.02 [-0.028 to -0.012]
Statistical Analysis 1: Comparison: Stable ICS-LABA vs Reduced ICS/LABA; Comparison of change in FEV1/FVC ratio; Test type: Superiority or Other; p = 0.14, Kruskal-Wallis
Statistical Analysis 2: Comparison: Stable ICS-LABA vs LABA Step Off; Comparison of change in FEV1/FVC ratio; Test type: Superiority or Other; p < 0.001, Kruskal-Wallis
Statistical Analysis 3: Comparison: Reduced ICS/LABA vs LABA Step Off; Comparison of change in FEV1/FVC ratio; Test type: Superiority or Other; p = 0.031, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: Adverse events were assessed via a questionnaire in the clinic visit form, which was completed at every visit. Adverse events were recorded for participants who had newly detected moderate or severe symptoms after baseline.
Arm/Group | Stable ICS-LABA | Reduced ICS/LABA | LABA Step Off
Serious Adverse Events (participants affected / at risk) | 7/151 | 3/149 | 15/155
Other Adverse Events (participants affected / at risk) | 110/151 | 102/149 | 100/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stable ICS-LABA (N=151) | Reduced ICS/LABA (N=149) | LABA Step Off (N=155)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort, shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stroke (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Acute renal failure, resolved (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Elevated blood sugar (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Graves' Disease, diagnosis (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Partial small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Appendectomy (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Knee replacement (planned) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Pregnancy (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 0 (0)
Hospitalized for contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stable ICS-LABA (N=151) | Reduced ICS/LABA (N=149) | LABA Step Off (N=155)
Skin bruising (Skin and subcutaneous tissue disorders) | 12 (12) | 8 (8) | 9 (9)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 45 (48) | 34 (35) | 46 (48)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 24 (28) | 35 (37) | 34 (35)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 26 (30) | 34 (34) | 21 (21)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 16 (16) | 18 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 53 (55) | 56 (59) | 58 (61)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 34 (36) | 23 (25) | 26 (27)
Headache (General disorders) | 38 (39) | 24 (29) | 37 (40)
Increased/irregular heartbeat (Cardiac disorders) | 6 (6) | 1 (1) | 6 (6)
Restlessness or nervousness (General disorders) | 17 (18) | 14 (15) | 13 (13)
Runny nose/congestion (Respiratory, thoracic and mediastinal disorders) | 52 (60) | 48 (58) | 52 (55)
Nausea/vomiting (Gastrointestinal disorders) | 16 (17) | 18 (18) | 12 (12)

LIMITATIONS AND CAVEATS:
At the time of this release, this data has not undergone peer-review.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No